CLINICAL TRIAL: NCT01642914
Title: Phase 3b, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Trial of Linaclotide Administered Orally for 12 Weeks to Patients With Chronic Constipation and Prominent Abdominal Bloating at Baseline
Brief Title: Safety and Efficacy of Linaclotide in Patients With Chronic Constipation and Prominent Abdominal Bloating
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIN-MD-04
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Constipation; Constipation
Keywords: Chronic Constipation; Abdominal Bloating; Linaclotide
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Linaclotide 290 micrograms (Experimental): Linaclotide 290 micrograms
  Interventions: Drug: Linaclotide 290 micrograms
- Linaclotide 145 Micrograms (Experimental): Linaclotide 145 micrograms
  Interventions: Drug: Linaclotide 145 micrograms
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Linaclotide 290 micrograms — oral capsule, taken once daily each morning at least 30 minutes before breakfast
  Arms: Linaclotide 290 micrograms
Drug: Linaclotide 145 micrograms — oral capsule, taken once daily each morning at least 30 minutes before breakfast
  Arms: Linaclotide 145 Micrograms
Drug: Matching placebo — oral capsule, taken once daily each morning at least 30 minutes before breakfast
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of linaclotide compared with placebo in patients with chronic constipation (CC) and prominent abdominal bloating. This study includes an up to 3-week screening period and a 2-3 week pretreatment period. Patients who are eligible will be randomized to one of two doses of linaclotide or placebo for 12 weeks. This 12-week study will assess the effects of linaclotide on bowel movement frequency, as well as other abdominal and bowel symptoms of CC.

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed a colonoscopy according to the American Gastroenterological Association criteria with no clinically significant findings
* Patient has successfully completed protocol procedures (with no clinically significant findings)
* Patient meets protocol criteria for Chronic Constipation(CC): < 3 bowel movements per week and reports one or more of the following symptoms for at least 12 weeks:

  1. Straining during more than 25% of BMs
  2. Lumpy or hard stools during more than 25% of BMs
  3. Sensation of incomplete evacuation during more than 25% of BMs
* Patient demonstrates continued chronic constipation and bloating through Pretreatment Period
* Patient is compliant with Interactive voice response System (IVRS)

Exclusion Criteria:

* Patient has a history of loose or watery stools
* Patient has symptoms of or been diagnosed with Irritable Bowel Syndrome (IBS)
* Patient has a structural abnormality of the gastrointestinal (GI) tract or a disease or condition that can affect GI motility
* Patient has any protocol-excluded or clinically significant medical or surgical history that would limit the patient's ability to complete or participate in this clinical trial or could confound the study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shiff, MD, Study Director — Forest Laboratories
Locations (151):
- United States (146):
  - Forest Investigative Site 020, Chandler, Arizona
  - Forest Investigative Site 102, Chandler, Arizona
  - Forest Investigative Site 149, Glendale, Arizona
  - Forest Investigative Site 126, Goodyear, Arizona
  - Forest Investigative Site 018, Phoenix, Arizona
  - Forest Investigative Site 061, Phoenix, Arizona
  - Forest Investigative Site 022, Scottsdale, Arizona
  - Forest Investigative Site 079, Tucson, Arizona
  - Forest Investigative Site 071, Tucson, Arizona
  - Forest Investigative Site 135, North Little Rock, Arkansas
  - Forest Investigative Site 106, Anaheim, California
  - Forest Investigative Site 104, Laguna Hills, California
  - Forest Investigative Site 066, Mission Hills, California
  - Forest Investigative Site 095, San Carlos, California
  - Forest Investigative Site 009, San Diego, California
  - Forest Investigative Site 151, Santa Monica, California
  - Forest Investigative Site 010, Westlake Village, California
  - Forest Investigative Site 012, Boulder, Colorado
  - Forest Investigative Site 041, Colorado Springs, Colorado
  - Forest Investigative Site 045, Colorado Springs, Colorado
  - Forest Investigative Site 060, Longmont, Colorado
  - Forest Investigative Site 007, Bristol, Connecticut
  - Forest Investigative Site 153, Waterbury, Connecticut
  - Forest Investigative Site 091, Boynton Beach, Florida
  - Forest Investigative Site 047, Bradenton, Florida
  - Forest Investigative Site 042, Brooksville, Florida
  - Forest Investigative Site 133, Coral Gables, Florida
  - Forest Investigative Site 131, DeLand, Florida
  - Forest Investigative Site 051, Fort Myers, Florida
  - Forest Investigative Site 137, Inverness, Florida
  - Forest Investigative Site 114, Jacksonville, Florida
  - Forest Investigative Site 004, Jupiter, Florida
  - Forest Investigative Site 016, Kissimmee, Florida
  - Forest Investigative Site 097, Lauderdale Lakes, Florida
  - Forest Investigative Site 003, Miami, Florida
  - Forest Investigative Site 002, Miami, Florida
  - Forest Investigative Site 130, New Smyrna Beach, Florida
  - Forest Investigative Site 040, Ocala, Florida
  - Forest Investigative Site 083, Orlando, Florida
  - Forest Investigative Site 150, Oviedo, Florida
  - Forest Investigative Site 132, Port Orange, Florida
  - Forest Investigative Site 127, Seminole, Florida
  - Forest Investigative Site 087, St. Petersburg, Florida
  - Forest Investigative Site 064, Tampa, Florida
  - Forest Investigative Site 115, Zephyrhills, Florida
  - Forest Investigative Site 021, Marietta, Georgia
  - Forest Investigative Site 011, Marietta, Georgia
  - Forest Investigative Site 109, Sandy Springs, Georgia
  - Forest Investigative Site 037, Stockbridge, Georgia
  - Forest Investigative Site 023, Woodstock, Georgia
  - Forest Investigative Site 015, Idaho Falls, Idaho
  - Forest Investigative Site 122, Peoria, Illinois
  - Forest Investigative Site 043, Rockford, Illinois
  - Forest Investigative Site 107, Anderson, Indiana
  - Forest Investigative Site 117, Clive, Iowa
  - Forest Investigative Site 146, Clive, Iowa
  - Forest Investigative Site 143, Davenport, Iowa
  - Forest Investigative Site 055, Iowa City, Iowa
  - Forest Investigative Site 028, Newton, Kansas
  - Forest Investigative Site 112, Overland Park, Kansas
  - Forest Investigative Site 034, Wichita, Kansas
  - Forest Investigative Site 032, Wichita, Kansas
  - Forest Investigative Site 128, Lexington, Kentucky
  - Forest Investigative Site 134, Madisonville, Kentucky
  - Forest Investigative Site 121, Baton Rouge, Louisiana
  - Forest Investigative Site 124, Metairie, Louisiana
  - Forest Investigative Site 101, Monroe, Louisiana
  - Forest Investigative Site 058, Shreveport, Louisiana
  - Forest Investigative Site 099, Shreveport, Louisiana
  - Forest Investigative Site 062, Baltimore, Maryland
  - Forest Investigative Site 008, Chevy Chase, Maryland
  - Forest Investigative Site 014, Hagerstown, Maryland
  - Forest Investigative Site 024, Towson, Maryland
  - Forest Investigative Site 006, Boston, Massachusetts
  - Forest Investigative Site 070, Chesterfield, Michigan
  - Forest Investigative Site 145, Traverse City, Michigan
  - Forest Investigative Site 141, Jackson, Mississippi
  - Forest Investigative Site 077, Fremont, Nebraska
  - Forest Investigative Site 048, Omaha, Nebraska
  - Forest Investigative Site 052, Henderson, Nevada
  - Forest Investigative Site 080, Las Vegas, Nevada
  - Forest Investigative Site 036, Clifton, New Jersey
  - Forest Investigative Site 088, Marlton, New Jersey
  - Forest Investigative Site 033, Vineland, New Jersey
  - Forest Investigative Site 063, Albuquerque, New Mexico
  - Forest Investigative Site 093, Albuquerque, New Mexico
  - Forest Investigative Site 044, Brooklyn, New York
  - Forest Investigative Site 017, Great Neck, New York
  - Forest Investigative Site 142, Asheboro, North Carolina
  - Forest Investigative Site 094, Asheville, North Carolina
  - Forest Investigative Site 075, Boone, North Carolina
  - Forest Investigative Site 123, Chapel Hill, North Carolina
  - Forest Investigative Site 140, Davidson, North Carolina
  - Forest Investigative Site 039, Fayetteville, North Carolina
  - Forest Investigative Site 031, Greensboro, North Carolina
  - Forest Investigative Site 029, Greensboro, North Carolina
  - Forest Investigative Site 078, Greensboro, North Carolina
  - Forest Investigative Site 084, Harrisburg, North Carolina
  - Forest Investigative Site 073, Hickory, North Carolina
  - Forest Investigative Site 050, Hickory, North Carolina
  - Forest Investigative Site 139, High Point, North Carolina
  - Forest Investigative Site 027, Raleigh, North Carolina
  - Forest Investigative Site 119, Statesville, North Carolina
  - Forest Investigative Site 089, Wilmington, North Carolina
  - Forest Investigative Site 074, Winston-Salem, North Carolina
  - Forest Investigative Site 025, Cincinnati, Ohio
  - Forest Investigative Site 120, Cincinnati, Ohio
  - Forest Investigative Site 056, Cleveland, Ohio
  - Forest Investigative Site 026, Columbus, Ohio
  - Forest Investigative Site 098, Dayton, Ohio
  - Forest Investigative Site 090, Dayton, Ohio
  - Forest Investigative Site 085, Mentor, Ohio
  - Forest Investigative Site 068, Wadsworth, Ohio
  - Forest Investigative Site 118, Oklahoma City, Oklahoma
  - Forest Investigative Site 081, Levittown, Pennsylvania
  - Forest Investigative Site 001, Pittsburgh, Pennsylvania
  - Forest Investigative Site 110, Reading, Pennsylvania
  - Forest Investigative Site 116, Greer, South Carolina
  - Forest Investigative Site 046, Simpsonville, South Carolina
  - Forest Investigative Site 092, Dakota Dunes, South Dakota
  - Forest Investigative Site 129, Chattanooga, Tennessee
  - Forest Investigative Site 138, Kingsport, Tennessee
  - Forest Investigative Site 125, Austin, Texas
  - Forest Investigative Site 035, Dallas, Texas
  - Forest Investigative Site 005, Dallas, Texas
  - Forest Investigative Site 111, Fort Worth, Texas
  - Forest Investigative Site 100, Houston, Texas
  - Forest Investigative Site 067, Katy, Texas
  - Forest Investigative Site 049, Pasadena, Texas
  - Forest Investigative Site 030, San Antonio, Texas
  - Forest Investigative Site 076, San Antonio, Texas
  - Forest Investigative Site 065, Sugarland, Texas
  - Forest Investigative Site 019, Ogden, Utah
  - Forest Investigative Site 105, Salt Lake City, Utah
  - Forest Investigative Site 113, Sandy City, Utah
  - Forest Investigative Site 053, Charlottesville, Virginia
  - Forest Investigative Site 108, Chesapeake, Virginia
  - Forest Investigative Site 136, Chesapeake, Virginia
  - Forest Investigative Site 148, Christiansburg, Virginia
  - Forest Investigative Site 072, Lynchburg, Virginia
  - Forest Investigative Site 069, Newport News, Virginia
  - Forest Investigative Site 013, Norfolk, Virginia
  - Forest Investigative Site 038, Richmond, Virginia
  - Forest Investigative Site 103, Spokane, Washington
  - Forest Investigative Site 082, La Crosse, Wisconsin
  - Forest Investigative Site 096, Milwaukee, Wisconsin
- Canada (5):
  - Forest Investigative Site 054, Greater Sudbury, Ontario
  - Forest Investigative Site 059, Sarnia, Ontario
  - Forest Investigative Site 086, Toronto, Ontario
  - Forest Investigative Site 147, Toronto, Ontario
  - Forest Investigative Site 152, Vaughan, Ontario

REFERENCES:
- [Derived] Lacy BE, Shea EP, Manuel M, Abel JL, Jiang H, Taylor DCA. Lessons learned: Chronic idiopathic constipation patient experiences with over-the-counter medications. PLoS One. 2021 Jan 11;16(1):e0243318. doi: 10.1371/journal.pone.0243318. eCollection 2021. PMID 33428631
- [Derived] Lacy BE, Schey R, Shiff SJ, Lavins BJ, Fox SM, Jia XD, Blakesley RE, Hao X, Cronin JA, Currie MG, Kurtz CB, Johnston JM, Lembo AJ. Linaclotide in Chronic Idiopathic Constipation Patients with Moderate to Severe Abdominal Bloating: A Randomized, Controlled Trial. PLoS One. 2015 Jul 29;10(7):e0134349. doi: 10.1371/journal.pone.0134349. eCollection 2015. PMID 26222318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred at 136 study sites in the US and 5 study sites in Canada over a 6 month period from August of 2012 to February of 2013.
Pre-assignment Details: Enrolled participants had up to 21 days of screening (screening period) to determine eligibility for entry into the study's pretreatment period. After an additional 14 to 21 days of pretreatment, those patients meeting entry criteria were randomized for 12 weeks of double-blind treatment.
Period: Overall Study
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Started | 173 | 154 | 160
Completed | 127 | 122 | 120
Not Completed | 46 | 32 | 40
Not completed — Adverse Event | 11 | 7 | 15
Not completed — Lack of Efficacy | 9 | 4 | 2
Not completed — Protocol Violation | 15 | 13 | 6
Not completed — Withdrawal by Subject | 5 | 5 | 10
Not completed — Lost to Follow-up | 5 | 3 | 7
Not completed — Other Reason | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 487 patients were randomized to treatment (Randomized Population). The Safety population consists of the 486 randomized who received at least one dose of study drug. The Demographic and Baseline Characteristics data reported here is for the Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms | Total
Number analyzed (Participants) | 173 | 153 | 160 | 486
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.3 (13.4) | 48.3 (12.6) | 47.5 (13.6) | 47.3 (13.2)
Age, Customized [Number; unit: participants]
  Age 18 to 39 years | 53 | 37 | 43 | 133
  Age 40 to 64 years | 104 | 104 | 99 | 307
  Age ≥ 65 years | 16 | 12 | 18 | 46
Sex/Gender, Customized [Number; unit: participants]
  Male | 14 | 15 | 12 | 41
  Female | 159 | 138 | 148 | 445
Race/Ethnicity, Customized [Number; unit: participants]
  White | 120 | 97 | 112 | 329
  Black or African American | 47 | 54 | 47 | 148
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 3 | 1 | 0 | 4
  Other | 3 | 1 | 0 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 26 | 19 | 25 | 70
  Non-Hispanic | 147 | 134 | 135 | 416
Region of Enrollment [Number; unit: participants]
  United States | 165 | 147 | 152 | 464
  Canada | 8 | 6 | 8 | 22
Weight, mean [Mean (Standard Deviation); unit: kg] | 77.59 (19.19) | 79.39 (18.01) | 80.53 (18.20) | 79.12 (18.50)
Height, mean [Mean (Standard Deviation); unit: cm] | 164.87 (8.65) | 164.85 (8.44) | 164.37 (7.07) | 164.70 (8.08)
BMI (Body Mass Index), mean [Mean (Standard Deviation); unit: kilograms per meter squared] | 28.43 (6.03) | 29.17 (6.03) | 29.83 (6.57) | 29.12 (6.23)

OUTCOME MEASURES:

1. Secondary Outcome: 9/12 Week Complete Spontaneous Bowel Movement (CSBM) 3+1 Responder
Description: A 9/12 Week CSBM 3+1 Responder is a patient who is a CSBM 3+1 Weekly Responder for at least 9 out of the 12 weeks of the Treatment Period. A CSBM 3+1 Weekly Responder is a patient who had a CSBM Weekly Frequency Rate that was 3 or greater and increased by 1 or more from baseline.
Time Frame: 12-week treatment period
Population: 487 patients were randomized to treatment (Randomized Population). The Safety population consists of 486 randomized patients who received at least one dose of study drug. The Intent to Treat (ITT) population consists of 483 patients in the Safety population with valid post-baseline efficacy data. Reported outcome data is based on the ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Linaclotide 290 Micrograms
Number analyzed (Participants) | 171 | 159
participants
  Responder | 13 | 26
  Nonresponder | 158 | 133

2. Secondary Outcome: Change From Baseline in 12-Week Abdominal Bloating
Description: Abdominal Bloating was measured daily using an 11-point Numerical Rating Scale (NRS) where a value of 0 represents no abdominal bloating and a value of 10 represents very severe abdominal bloating. The abdominal bloating score from Baseline is derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization up to the time of randomization (Visit 3, Day 1). The change from baseline in 12-Week Abdominal Bloating score is the difference between the average nonmissing daily patient assessments of abdominal bloating scores during the 14 day Baseline period, and the average of the nonmissing daily patient assessments of abdominal bloating scores reported during the 12 week Treatment Period.
Time Frame: Baseline and 12-week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 171 | 153 | 159
units on a scale | -1.583 (1.988) | -2.476 (2.315) | -2.456 (2.240)

3. Secondary Outcome: Percent Change From Baseline in 12-week Abdominal Bloating
Description: Abdominal Bloating was measured daily using an 11-point Numerical Rating Scale (NRS) where a value of 0 represents no abdominal bloating and a value of 10 represents very severe abdominal bloating. The abdominal bloating score from Baseline is derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). The percent change from baseline in 12-Week Abdominal Bloating score is the percentage difference between the average nonmissing daily patient assessments score of abdominal bloating scores during the 14 day Baseline period, and the average of the nonmissing daily patient assessments of abdominal bloating scores reported during the 12 week Treatment Period.
Time Frame: Baseline and 12-week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change of NRS score
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 171 | 153 | 159
percentage change of NRS score | -22.65 (29.19) | -34.52 (31.79) | -34.22 (30.65)

4. Secondary Outcome: Percent Change From Baseline in Abdominal Bloating at Week 12
Description: Abdominal bloating was measured daily using an 11-point Numerical Rating Scale (NRS) where a value of 0 represents no abdominal bloating and a value of 10 represents very severe abdominal bloating. The abdominal bloating score from Baseline is derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). The percent change from baseline at Week 12 in Abdominal Bloating score is the percentage difference between the average nonmissing daily patient assessments of abdominal bloating scores during the 14 day Baseline period, and the average of the nonmissing daily patient assessments of abdominal bloating scores reported during Week 12.
Time Frame: Baseline and Week 12
Population: Reported outcome data is based on the 483 patient Intent-to-Treat Population. The distribution of each of the linaclotide groups was compared, in a pair-wise manner, to the placebo group using the two-sample Kolmogorov-Smirnov test.
Measure: Mean (Standard Deviation); unit: percentage change in abdominal bloating
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 135 | 121 | 118
percentage change in abdominal bloating | -31.41 (40.78) | -45.43 (37.56) | -47.12 (33.55)
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 145 Micrograms; Test type: Superiority or Other; p = 0.0054, Kolmogorov-Smirnov; Kolmogorov-Smirnov test for equality of distribution
Statistical Analysis 2: Comparison: Placebo vs Linaclotide 290 Micrograms; Test type: Superiority or Other; p = 0.0012, Kolmogorov-Smirnov; Kolmogorov-Smirnov test for equality of distribution

5. Secondary Outcome: 6/12 Week Abdominal Bloating 30% Responder
Description: A patient was a 6/12 week abdominal bloating 30% responder if, for at least 6 weeks of the 12-week treatment period, that patient's improvement from baseline in the weekly abdominal bloating score was ≥ 30% from baseline.
Time Frame: 12-week treatment period
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 171 | 153 | 159
participants
  Responder | 50 | 62 | 69
  Nonresponder | 121 | 91 | 90

6. Secondary Outcome: Change From Baseline in 12-week CSBM Frequency Rate
Description: A patient's 12-week CSBM frequency rate from Baseline is derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). A patient's 12-week CSBM frequency rate was the CSBM rate (CSBMs/week) calculated over the 12 weeks of the treatment period.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: Baseline and 12-week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CSBMs per week
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 171 | 153 | 159
CSBMs per week | 1.020 (1.596) | 2.309 (2.832) | 2.292 (2.790)

7. Secondary Outcome: Change From Baseline in CSBM Frequency Rate at Week 1.
Description: A patient's CSBM frequency rate from Baseline is derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). A patient's CSBM frequency rate at week 1 was the CSBM rate (CSBMs/week) calculated over that week.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CSBMs per week
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 171 | 153 | 159
CSBMs per week | 0.641 (1.543) | 1.984 (3.784) | 1.746 (2.842)

8. Secondary Outcome: Change From Baseline in CSBM Frequency Rate at Week 4.
Description: A patient's CSBM frequency rate from Baseline is derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). A patient's CSBM frequency rate at week 4 was the CSBM rate (CSBMs/week) calculated over that week.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CSBMs per week
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 164 | 144 | 145
CSBMs per week | 1.063 (2.176) | 2.756 (3.662) | 2.678 (3.552)

9. Secondary Outcome: Change From Baseline in CSBM Frequency Rate at Week 8
Description: A patient's CSBM frequency rate from Baseline is derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). A patient's CSBM frequency rate at week 8 was the CSBM rate (CSBMs/week) calculated over that week.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CSBMs per week
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 147 | 133 | 131
CSBMs per week | 1.347 (2.438) | 2.803 (4.034) | 2.319 (2.989)

10. Secondary Outcome: Change From Baseline in CSBM Frequency Rate at Week 12
Description: A patient's CSBM frequency rate from Baseline is derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). A patient's CSBM frequency rate at week 12 was the CSBM rate (CSBMs/week) calculated over that week.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CSBMs per week
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 137 | 126 | 124
CSBMs per week | 1.074 (1.893) | 2.272 (2.801) | 2.488 (3.010)

11. Secondary Outcome: Change From Baseline in 12-Week SBM Frequency Rate
Description: A patient's Baseline SBM frequency rate is derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). A patient's 12-week SBM frequency rate was the SBM rate (SBMs/week) calculated over the 12 weeks of the treatment period.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: 12-week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SBMs per week
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 171 | 153 | 159
SBMs per week | 1.480 (2.198) | 3.481 (3.085) | 3.550 (3.382)

12. Secondary Outcome: Change From Baseline in SBM Frequency Rate at Week 1
Description: A patient's baseline SBM frequency rate is derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). A patient's SBM frequency rate at week 1 was the SBM rate (SBMs/week) calculated over that week.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SBMs per week
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 171 | 153 | 159
SBMs per week | 1.840 (2.520) | 4.168 (4.547) | 4.125 (4.229)

13. Secondary Outcome: Change From Baseline in SBM Frequency Rate at Week 4
Description: A patient's baseline SBM frequency rate is derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). A patient's SBM frequency rate at Week 4 was the SBM rate (SBMs/week) calculated over that week.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SBMs per week
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 164 | 144 | 145
SBMs per week | 1.420 (2.882) | 4.045 (4.172) | 3.872 (4.563)

14. Secondary Outcome: Change From Baseline in SBM Frequency Rate at Week 8
Description: A patient's baseline SBM frequency rate is derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). A patient's SBM frequency rate at Week 8 was the SBM rate (SBMs/week) calculated over that week.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SBMs per week
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 147 | 133 | 131
SBMs per week | 1.638 (3.093) | 3.674 (3.784) | 3.785 (3.925)

15. Secondary Outcome: Change From Baseline in SBM Frequency Rate at Week 12
Description: A patient's baseline SBM frequency rate is derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). A patient's SBM frequency rate at week 12 was the SBM rate (SBMs/week) calculated over that week.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SBMs per week
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 137 | 126 | 124
SBMs per week | 1.288 (2.221) | 3.085 (3.399) | 2.983 (3.616)

16. Secondary Outcome: Change From Baseline in the Number of Days With a Spontaneous Bowel Movement (SBM)
Description: A patient's baseline number of days with a Spontaneous Bowel Movement (SBM) was calculated as the number of days with at least 1 Spontaneous Bowel Movement (SBM), derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). A patient's number of days with a SBM during the Treatment Period was calculated as the number of days with at least 1 Spontaneous Bowel Movement (SBM), divided by treatment duration (in days), and multiplied by 7.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: Baseline and 12-week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days per week
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 171 | 153 | 159
Days per week | 1.086 (1.595) | 2.279 (1.830) | 2.143 (1.780)

17. Secondary Outcome: SBM Within 24 Hours After the First Dose of Investigational Product
Description: The proportion of patients with a SBM within 24 hours of first taking investigational product in each linaclotide dose group was compared with the proportion in the placebo group using the Cochran-Mantel-Haenszel (CMH) test controlling for geographic region.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: 24 hours from first dose of investigational product (Day 1)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 171 | 153 | 159
participants
  Responder | 72 | 94 | 94
  Nonresponder | 99 | 59 | 65
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 145 Micrograms; Test type: Superiority or Other; p = 0.0006, Cochran-Mantel-Haenszel — p-Values were obtained from the Cochran-Mantel-Haenszel tests controlling for geographic region, comparing each linaclotide dose versus placebo in a pairwise manner; Risk Difference (RD) = .193, 95% CI 2-sided [.086 to .300]
Statistical Analysis 2: Comparison: Placebo vs Linaclotide 290 Micrograms; Test type: Superiority or Other; p = 0.0022, Cochran-Mantel-Haenszel — [p-value comment as in outcome 17, analysis 1]; Risk Difference (RD) = .170, 95% CI 2-sided [.064 to .227]

18. Secondary Outcome: Time to Spontaneous Bowel Movement (SBM) After the First Dose of Investigational Product
Description: Time to first SBM after the first dose of investigation product was defined as the number of hours between the time of the first dose of investigational product to the occurrence of the first SBM. Patients who did not achieve an SBM were considered censored, with time to censoring defined as the number of hours elapsing from the time of the first dose of investigational product was taken to the end of the day of the last dose, at 12:00 AM (24:00 military time).
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: 12-week treatment period
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 171 | 153 | 159
Hours | 28.07 [24.02 to 43.27] | 12.53 [7.03 to 21.18] | 19.35 [9.81 to 23.02]
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 145 Micrograms; Test type: Superiority or Other; p = .0054, Log Rank; Log-rank test stratified by geographic region; Cox Proportional Hazard = 1.37, 95% CI 2-sided [1.09 to 1.72]
Statistical Analysis 2: Comparison: Placebo vs Linaclotide 290 Micrograms; Test type: Superiority or Other; p = 0.0470, Log Rank; Log-rank test stratified by geographic region; Cox Proportional Hazard = 1.24, 95% CI 2-sided [0.99 to 1.55]

19. Secondary Outcome: Change From Baseline in 12-week Stool Consistency
Description: Stool consistency was measured using the 7-point Bristol Stool Form Scale (BSFS):
  1. = separate hard lumps like nuts [difficult to pass]
  2. = sausage shaped but lumpy
  3. = like a sausage but with cracks on surface
  4. = like a sausage or snake, smooth and soft
  5. = soft blobs with clear-cut edges [passed easily]
  6. = fluffy pieces with ragged edges, a mushy stool
  7. = watery, no solid pieces [entirely liquid]
  A patient's BSFS score for the baseline period (14 days before randomization, up to the time of randomization) and for the 12-week treatment period, was the average of the nonmissing BSFS scores from the SBMs reported by the patient during the respective baseline and treatment periods.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: Baseline and 12-week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 160 | 137 | 137
units on a scale | 0.797 (1.129) | 1.925 (1.358) | 2.304 (1.470)

20. Secondary Outcome: Change From Baseline in Stool Consistency at Week 12
Description: Stool consistency was measured using the 7-point Bristol Stool Form Scale (BSFS):
  1. = separate hard lumps like nuts [difficult to pass]
  2. = sausage shaped but lumpy
  3. = like a sausage but with cracks on surface
  4. = like a sausage or snake, smooth and soft
  5. = soft blobs with clear-cut edges [passed easily]
  6. = fluffy pieces with ragged edges, a mushy stool
  7. = watery, no solid pieces [entirely liquid]
  A patient's BSFS score for the baseline period (14 days before randomization, up to the time of randomization) and at week 12, was the average of the nonmissing BSFS scores from the SBMs reported by the patient during the respective baseline period and during Week 12.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 116 | 105 | 99
units on a scale | 0.845 (1.439) | 2.061 (1.478) | 2.358 (1.687)

21. Secondary Outcome: Change From Baseline in 12-week Severity of Straining
Description: Severity of straining was measured using a 5-point ordinal scale, where of value of 1 is "not at all" and a value of 5 is "an extreme amount." A patient's straining score for baseline was derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). A patient's straining score for the treatment period was the average of the nonmissing straining scores from the SBMs reported by the patient during the 12-week treatment period.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: Baseline and 12-week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 160 | 136 | 137
units on a scale | -0.812 (0.941) | -1.495 (0.938) | -1.512 (1.027)

22. Secondary Outcome: Change From Baseline in Severity of Straining at Week 12
Description: Severity of straining was measured using a 5-point ordinal scale, where of value of 1 is "not at all" and a value of 5 is "an extreme amount."
  A patient's straining score for baseline was derived from the Interactive Voice Response System (IVRS) daily diary data collected in the Pretreatment Period, specifically the period of time from 14 days before randomization, up to the time of randomization (Visit 3, Day 1). A patient's straining score at Week 12 was the average of the nonmissing straining scores from the SBMs reported by that patient during analysis Week 12.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 116 | 105 | 99
units on a scale | -1.021 (1.184) | -1.654 (0.970) | -1.686 (1.117)

23. Secondary Outcome: 9/12 Week Mild Straining and Diarrhea-free Responder
Description: A patient was a 9/12 week mild straining and diarrhea-free responder if that patient met the weekly criterion for at least 9 weeks of the 12-week treatment period. A patient was considered to have met the weekly criterion in a given week if that patient had a nonmissing average straining score ≤ 2 (where a value of 1 represents no straining, an a value of 5 represents an extreme amount of straining), and the patient had no diarrhea adverse event (AE) reported for that week.
  Only the Placebo versus Linaclotide 145 micrograms arm comparison is a secondary measure type for this outcome measure. The additional data for the Linaclotide 290 micrograms arm (a pre-specified additional outcome measure) is presented here for ease of comparison.
Time Frame: 12-week treatment period
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Number analyzed (Participants) | 171 | 153 | 159
participants
  Responder | 15 | 38 | 27
  Nonresponder | 156 | 115 | 132

24. Primary Outcome: 9/12 Week Complete Spontaneous Bowel Movement (CSBM) 3+1 Responder
Description: as for outcome 1
Time Frame: 12-week treatment period
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Linaclotide 145 Micrograms
Number analyzed (Participants) | 171 | 153
participants
  Responder | 13 | 24
  Nonresponder | 158 | 129
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 145 Micrograms; Test type: Superiority or Other; p = 0.0264, Cochran-Mantel-Haenszel — [p-value comment as in outcome 17, analysis 1]; Odds Ratio (OR) = 2.23, 95% CI 2-sided [1.09 to 4.56]

ADVERSE EVENTS:
Time Frame: Adverse event reporting occurred over a 10 month period from August of 2012 to June of 2013 at 141 study sites in the United States and Canada
Arm/Group | Placebo | Linaclotide 145 Micrograms | Linaclotide 290 Micrograms
Serious Adverse Events (participants affected / at risk) | 2/173 | 4/153 | 2/160
Other Adverse Events (participants affected / at risk) | 12/173 | 25/153 | 33/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=173) | Linaclotide 145 Micrograms (N=153) | Linaclotide 290 Micrograms (N=160)
brain stem infarction (Nervous system disorders) | 1 | 0 | 0
abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
non-cardiac chest pain (General disorders) | 0 | 1 | 0
gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
pneumonia (Infections and infestations) | 0 | 0 | 1
anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=173) | Linaclotide 145 Micrograms (N=153) | Linaclotide 290 Micrograms (N=160)
Diarrhoea (Gastrointestinal disorders) | 4 | 9 | 27
Upper respiratory tract infection (Infections and infestations) | 5 | 9 | 5
Sinusitis (Infections and infestations) | 3 | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this trial will be the property of Forest Research Institute, Inc. and Ironwood Pharmaceuticals, Inc. An integrated clinical and statistical report will be prepared at the completion of the trial.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator, Ironwood Pharmaceuticals, Inc., and Forest Research Institute, Inc.